CLINICAL TRIAL: NCT03620370
Title: The Safety and Efficacy of Normobaric Hyperoxia Combined With Reperfusion for Acute Ischemic Stroke：A Randomized, Controlled Pilot Study
Brief Title: Normobaric Hyperoxia Combined With Reperfusion for Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPENS-1
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2020-07

CONDITIONS: Stroke, Acute
Keywords: Normobaric hyperoxia;; Acute ischemic stroke;; vascular recanalization;; Endovascular treatment;; reperfusion therapy
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBO group (Experimental): Normobaric oxygen therapy is the delivery of high-flow oxygen (10L/min) via oxygen storage facemask. This therapy should start in the pre-hospital or emergency room as soon as possible (within 1 hours) after diagnosis of ischemic stroke and last for 4 hours. All participant will receive mechanical thrombectomy and a standard clinical therapy.
  Interventions: Drug: Normobaric oxygen therapy
- Control group (No Intervention): The participants receive mechanical thrombectomy therapy after diagnosed ischemic. All participants receive a standard clinical therapy.

INTERVENTIONS:
Drug: Normobaric oxygen therapy — In this study, it is simple to administer via oxygen storage facemask at flow rates of 10 L/min for 4 hours. This therapy start should in Pre-hospital or emergency room as early as possible after diagnosed ischemic stroke and uninterrupted during other treatments including mechanical thrombolytic therapy and standard clinical treatment.
  Arms: NBO group

SUMMARY:
NBO is a nonpharmacological measure of neuroprotection. The purpose of our study is to evaluate the safety and efficiency of NBO（Normobaric hyperoxia) in the acute ischemic stroke patients who received endovascular treatment. Looking for more clinical evidence for the ischemic stroke patients who will be treated with NBO in the future.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age≥18 and ≤ 80;
* Suspected lage vessel occlusion of acute anterior circulation occlusion; i.e. either the ICA or the M1-segment of the MCA;
* Acute ischemic stroke where patient is ineligible for intravenous thrombolytic treatment or the treatment is contraindicated, or where patient has received intravenous thrombolytic therapy without recanalization;
* Patient treatable within 6 hours of symptom onset;or it has been more than 6 hours but not more than 24 hours,and imaging confirmed the existence of ischemic penumbra;
* NIHSS score≥6分
* Alberta Stroke Program Early CT score (ASPECTS) of 7-10 on non-contrast CT;
* Informed consent obtained;

Exclusion Criteria:

* Rapid improvement in neurological status to an NIHSS < 6 or evidence of vessel recanalization prior to randomization;
* Seizures at stroke onset;
* Intracranial hemorrhage;
* Systolic pressure greater than 185 mm Hg or diastolic pressure greater than 110 mm Hg, or aggressive treatment intravenous medication)necessary to reduce blood pressure to these limits;
* Symptoms rapidly improving;
* Symptoms suggestive of subarachnoid hemorrhage, even if CT scan was normal;
* Platelet count of less than 100,000 per cubic millimeter;
* CT showed a multiple infarction (low density area greater than 1/3 cerebral hemisphere);
* severe hepatic or renal dysfunction;
* active and chronic obstructive pulmonary disease or acute respiratory distress syndrome;
* >3 L/min oxygen required to maintain peripheral arterial oxygen saturation (SaO2)﹥95% as per current stroke management guidelines;
* medically unstable;
* inability to obtain informed consent;
* Life expectancy<90 days;
* Pregnant or breast-feeding women;
* Unwilling to be followed up or poor compliance for treatment;
* Patients being enrolled or having been enrolled in other clinical trial within 3 months prior to this clinical trial;
* Evidence of intracranial tumor;
* Baseline blood glucose of < 50 mg/dL (2.78 mmol) or > 400 mg/dL (22.20 mmol);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-08-12 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-10-19 (Actual)

PRIMARY OUTCOMES:
Cerebral infarct volume | 24-48h after randomization
  Infarct volume is evaluated mainly through brain MRI(DWI)

SECONDARY OUTCOMES:
levels of blood biomarkers | baseline; 24 ± 6 hours, 7 ± 2 days
  Biomarkers for evaluation of BBB damage and brain injury:NSE、S100B、occludin、 claudin-5、MMP-9
modified Rankin Scale score (mRS) | 30 ± 5 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint;the mRs is an ordinal disability score of 7 categories (0 = no symptoms to 5 = severe disability, and 6 = death)
The good prognosis at 90 days assessed by modified Rankin scale (mRS). | 90 ± 10 days after randomization
  secondary clinical efficacy endpoint;the mRs is an ordinal disability score of 7 categories (0 = no symptoms to 5 = severe disability, and 6 = death);The ratio of 0 to 2;
Scores assessed by National Institutes of Health Stroke Scale(NIHSS) | 2 hours ± 15 minutes, 24 ± 6 hours, 7 ± 2 days, 30 ± 5 days after randomization ]
  secondary clinical efficacy endpoint; the NIHSS is a stroke severity score that is composed of 11 items; range from 0 to 42, higher values indicate more severe deficits
Change in National Institutes of Health Stroke Scale (NIHSS) score from baseline to 24 hours | from baseline to 24 ± 6 hours
  secondary clinical efficacy endpoint;the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits)
Improvement of neurologic function after 24h | 24 ± 6 hours;
  NIHSS score decreased by more than 4 points or NIHSS score was 0;secondary clinical efficacy endpoint;the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits)
Barthel Index (BI) | 30 ± 5 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint;the BI is an ordinal disability score of 10 categories(range from 0 to 100, higher values indicate better prognosis);
Revascularization on 24-hour follow-up imaging | 24 (12 to 36) hours;
  secondary imaging efficacy endpoint;
24-hour neurologic deterioration; | 24 ± 6 hours;
  NIHSS score increased by more than 4 points);the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits);clinical safety endpoint;
any intracranial hemorrhage on 24-hour follow-up imaging | 24 (12 to 36) hours
  imaging safety endpoints;per ECASS III definition and per Heidelberg bleeding classification
Symptomatic Intracerebral Hemorrhage | 24 (12 to 36) hours
  imaging safety endpoints;Deterioration in NIHSS score of ≥4 points within 24 hours;per ECASS III definition and per Heidelberg bleeding classification
Mortality and Stroke recurrence | 90 ± 10 days after randomization
  clinical safety endpoint;
Survival rates | 7 ± 2 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint;
TICI (Thrombolysis in Cerebral Infarction perfusion scale grade) | Time Frame: 4 hours ± 15 minutes
  secondary imaging efficacy endpoint;
The infarct volume on 24-hour follow-up imaging | 24 (12 to 36) hours;
  The infarct volume of cerebral infarct is evaluated by cranial CT;
mRS4-6 | 90 ± 10 days after randomization
  secondary clinical efficacy endpoint;the mRs is an ordinal disability score of 7 categories (0 = no symptoms to 5 = severe disability, and 6 = death)

OTHER OUTCOMES:
Subgroup analysis of infarct volume | 24-48h after randomization
  Stratify according to different risk factors：ASPECT; NIHSS; age;Ischemic penumbra volume; Site of occlusion; Time from stroke onset to randomization;Ischemic penumbra volume

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu hospital;Capital Medical University, Beijin, China

REFERENCES:
- [Derived] Niu H, Ding J, Chen Z, Yuan S, Qi Z, Ji X, Li W. Normobaric Hyperoxia in Patients With Acute Stroke: Enhancing Neuroprotection Through Inhibition of Inflammation. J Am Heart Assoc. 2025 Oct 9:e041825. doi: 10.1161/JAHA.125.041825. Online ahead of print. PMID 41065265
- [Derived] Li W, Qi Z, Ma Q, Ding J, Wu C, Song H, Yang Q, Duan J, Liu L, Kang H, Wu L, Ji K, Zhao W, Li C, Sun C, Li N, Fisher M, Ji X, Liu KJ. Normobaric Hyperoxia Combined With Endovascular Treatment for Patients With Acute Ischemic Stroke: A Randomized Controlled Clinical Trial. Neurology. 2022 Aug 23;99(8):e824-e834. doi: 10.1212/WNL.0000000000200775. Epub 2022 Jun 17. PMID 35715198